CLINICAL TRIAL: NCT04923308
Title: The Effect of Chiropractor-informed Triage Versus Usual Medical Management on Low Back Pain Patient Outcomes and Trajectories in Tertiary Care Settings: a Controlled Clinical Study.
Brief Title: The Effect of Chiropractor-informed Triage on Low Back Pain Patient Outcomes and Trajectories
Status: Completed | Type: Observational
Sponsor: Université du Québec à Trois-Rivières (Other)
Responsible Party: Principal Investigator, Martin Descarreaux, Full professor, Université du Québec à Trois-Rivières
Other Study IDs: UQTR-2021-triage
Record Dates: First submitted 2021-06-02; First posted 2021-06-11 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Low Back Pain; Triage
Keywords: Low back pain; triage; care pathways; chiropractor; pain; disability; health resources
MeSH Terms: conditions — Low Back Pain; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Intervention group
  Interventions: Other: Triage results disclosed
- Control group
  Interventions: Other: Triage results undisclosed

INTERVENTIONS:
Other: Triage results disclosed — Following the chiropractor triage assessment, the working diagnosis and risk stratification or referral need will be communicated to the specialist using a standardized clinical note, prior to the patient's consultation and without further discussion.
  Groups: Intervention group
Other: Triage results undisclosed — Following the chiropractor triage assessment, the working diagnosis and risk stratification or referral need will not be communicated to the specialist.
  Groups: Control group

SUMMARY:
Almost everyone will have low back pain (LBP) at some point in their lives. LBP is a complex multifactorial condition for which diagnosis and clinical management remains a challenge. Factors such as wait times, delays in diagnosis or proper referral can result in Canadian patients having difficulty getting the care that they need. The overall objective of this project is to explore how chiropractors, who specialize in the diagnosis and clinical management of spinal conditions, can transform healthcare trajectories and improve the health of patients with LBP by integrating medical specialist team.To do so, patients with low back pain seeking medical care within the public health system will be first seen by chiropractors. Chiropractors will play a key role in identifying the type of low back pain and subsequently offering guidance to medical specialists with regard to the best treatment and management options that are currently recommended. Participating patients will be followed over a year while extensive health-related data will be collected and compared to non-triage patients with LBP.

ELIGIBILITY:
Inclusion Criteria:

* Being ≥ 18 years of age
* Being scheduled in the outpatient clinics with a primary complaint of LBP (either acute, chronic or recurring episodes), consistent with LBP definition (pain between the lower rib margins and the buttock creases, with or without associated symptoms in the lower limb(s)).
* Being able to comprehend and express oneself in French

Exclusion Criteria:

* Patients involved in litigation related to their LBP condition (i.e., worker's compensation, public automobile insurance plan or other litigations)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will involve individuals seeking medical consultation in the tertiary care public health system for an episode of LBP. The study will be conducted at the neurosurgery outpatient clinic affiliated to the Centre Intégré Universitaire de Santé et de Services Sociaux- Mauricie Centre du Québec (CIUSSS-MCQ; Trois-Rivières' regional healthcare organization). The CIUSSS-MCQ, established in 2015 as a result of the merger of 12 health and social services public institutions, totals 974 physicians, including 515 GPs. It serves a population of over 510,000 inhabitants, of which 83% are over 18 years of age (17).
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-11-27 (Actual)

PRIMARY OUTCOMES:
Change from baseline in back and leg pain intensity (current and past week) | baseline, week 1, week 12, week 24 and 12 months follow-up
  11-point numerical rating scale (NRS) :global measure of pain intensity anchored by two extremes of pain intensity ranging from 0 ('no pain') to 10 ('pain as bad as it could be').

SECONDARY OUTCOMES:
Diagnosis made by the specialist | up to 4 weeks post-baseline assessment
  The diagnosis and clinical management (i.e. self-management; including advice or brief intervention/medication), referral to other first line care practitioner (chiropractor, physiotherapist, etc.) or medical specialist, injection, leave of absence, etc.) decided by the specialist will be retrieved immediately after the initial encounter and compared to the chiropractor's working diagnosis, risk stratification or referral need according to current evidenced-bases practice guidelines
Number of requests for medical imaging | over a one year period
  Will be monitored through the patient's electronic clinical record (ECR), which is used in all health and social services across the Centre intégré universitaire de santé et de services sociaux de la Mauricie-et-du-Centre-du-Québec (CIUSSS-MCQ) institutions.
Number of requests for laboratory tests | over a one year period
  Will be monitored through the patient's electronic clinical record (ECR), which is used in all health and social services across the CIUSSS-MCQ institutions.
Number of requests for medication prescriptions | over a one year period
  Will be monitored through the patient's electronic clinical record (ECR), which is used in all health and social services across the CIUSSS-MCQ institutions.
Number of subsequent visits to the outpatient clinic or medical specialist | over a one year period
  Will be monitored (including date of visit, type of professional, number of visit, prescribe medication, referrals) through the patient's electronic clinical record (ECR), which is used in all health and social services across the CIUSSS-MCQ institutions.
Number of visit to non-publicity funded care | over a one year period
  Non-publicity funded care include any care that was fully paid out of pocket or reimbursed by a personal insurance coverage. This will be tracked by asking patients at follow-up if they sought first line care for their current LBP episode since the last assessment time point.
Disability | baseline, week 1, week 12, week 24 and 12 months follow-up
  Oswestry Disability Index (ODI): regroups ten questions related to different domains including pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sexual life, social life, and traveling. Each question is rated on a scale of 0 to 5 points with a maximum score of 50. Higher scores indicate greater disability
Number of significant pain episodes of LBP | over a one year period
  Defined as LBP episode lasting more than 24 h, preceded and separated by a period of at least 1 month without LBP; will be tracked with a personal diary.
Change from baseline Health-related quality of life | baseline, week 1, week 12, week 24 and 12 months follow-up
  WHO Quality of Life-BREF questionnaire: assesses the individual's perceptions in the context of their culture and value systems, and their personal goals, standards and concerns. The instrument comprises 26 items, which measure the following four domains: physical health, psychological health, social relationships, and environment. Higher scores denote higher quality of life
General expectations of recovery | baseline
  11-point NRS for which the patients will be asked the following question: How likely do you think it is that you will have a complete recovery? Possible answers ranging from -5= "very unlikely" to +5="very likely", with 0 being "I don't know''
Perceived Global Rating of Change | week 1, week 12, week 24 and 12 months follow-up
  Will be measured using the following question: With respect to your low back pain, how would you describe yourself now compared to the initial onset of symptoms? Participants will select between one of the seven following choices: 1) completely better; 2) much improved; 3) slightly improved; 4) no change; 5) slightly worse; 6) much worse and 7) worse than ever
Patient satisfaction | After the baseline assessment
  Patients will be asked to rate their experience with the chiropractor on a 5-point Likert scale (0=poor to 5=excellent) for each of the following items: 5-Time spent with the healthcare professional you saw; 6-Explanation of what was done for you; 7-Technical skills (thoroughness, carefulness, competence) of the healthcare professional you saw; 8-The personal (courtesy, respect, sensitivity, friendliness) of the person you saw; 9-The visit overall.

CONTACTS AND LOCATIONS:
Locations (1):
- Université du Québec à Trois-Rivières, Trois-Rivières, Quebec, Canada